CLINICAL TRIAL: NCT02695706
Title: Clinical Study, Opened, of Cutaneous Acceptability of a Topic Product in Normal Conditions of Use and Evaluation of the Effectiveness Through the Self Awareness of the Research, of Clinical Evaluations and Instrumental Measurements
Brief Title: Clinical Study, Opened, of Cutaneous Acceptability of a Topic Product in Normal Conditions of Use
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LM Farma Indústria e Comércio Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LM Farma
Record Dates: First submitted 2016-02-12; First posted 2016-03-01 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes
Keywords: Diabetes; Skin acceptability; Clinical Research
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laboratoires Mercurochrome Reparador (Experimental): A group of patients will be treated with a new restorative skin cream consists of hyperoxygenation essential fatty acids (60% linoleic acid) which does not contain preservatives (parabens) or known allergens.
  Interventions: Device: Laboratoires Mercurochrome Reparador

INTERVENTIONS:
Device: Laboratoires Mercurochrome Reparador — Developed for the treatment of damaged or fragile skin.
  Other Names: Urgo Repair

SUMMARY:
The measured product in this research is a product for topical use, Laboratoires Mercurochrome Reparador e Protetor. The expected benefit to the use of the product is the improvement in skin hydration as measured by self perception of participant research and clinical evaluation and improvement in local microcirculation, assessed by instrumental measurements in feet of the study participants.

DETAILED DESCRIPTION:
The objectives of this study is to verify the skin acceptability through the non-occurrence of adverse events and cutaneous sensations of discomfort, evaluate the moisturizing efficacy of the product through self perception of research participants and dermatological clinical evaluation to assess the improvement in local microcirculation by performing of instrumental measurements in the feet of diabetic participants, product Laboratoires Mercurochrome Repairer and Protector referred by LM FARMA INDUSTRIAL LTDA.

For this research, will be recruited up to 35 research participants who meet the inclusion / exclusion described in items 9.4 and 9.5 of the research protocol, to achieve a number of completion of 30 participants. Be recruited participants from both sexes, aged 18 and 65, which have dry skin on the feet and they are people with diabetes whose condition is stabilized.

ELIGIBILITY:
Inclusion Criteria:

* Participants healthy research;
* Intact skin on feet - grade 0 in the Wagner scale;
* Agreement to adhere to the procedures and requirements of the study and attend to the Office (s) day (s) and time (s) set (s) for evaluations;
* Ability to consent to participate in writing;
* Age 18 to 65 years;
* Research Participants of both sexes - including at least three men;
* Introducing dry skin on feet - dermatological proof.
* Participants with diabetes whose condition is stabilized

Exclusion Criteria:

* Pregnancy and lactation; skin pathology in the product application area;
* immune impairment;
* Current use of these medications for topical or systemic use: corticoid, immunosuppressants, antihistamines, anticoagulants or birth;
* Skin diseases: psoriasis, vitiligo, atopic dermatitis;
* History of reaction to the category of the product tested;
* Other diseases or medications that may interfere directly in the study or to endanger the health of the research participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Skin acceptability through the self perception of patients. | 2 months
  Measure the skin acceptability through the self perception of patients with the daily use of the product adding in a questionnaire the product effectiveness.

SECONDARY OUTCOMES:
Instrumental Performance Measures | 2 months
  Instrumental measurements will be carried out through the Skin-Thermometer ST equipment 500 - Courage + Khazaka in the feet of participants with the aid of a dermatologist.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Tepas, Graduated, Study Director — Urgo

IPD SHARING:
Plan to Share IPD: Undecided